CLINICAL TRIAL: NCT02890797
Title: Evaluation of Thoracic Echography for Pleuroparenchymatous Anomaly Diagnosis Complicating Bronchiolitis: BronchioIUS
Brief Title: Assessment of Thoracic Echography for Pleuroparenchymatous Anomaly Diagnosis Complicating Bronchiolitis: BronchioIUS
Acronym: BronchioIUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The inclusions have been suspended from 03/18/2020 during the confinement period.
  In the meantime, a publication has appeared showing that the chest ultrasound has entered the common practice in the management of bronchiolitis.
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/15/7858
Record Dates: First submitted 2016-07-12; First posted 2016-09-07 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; parenchymal condensation; chest X-ray; chest ultrasound
MeSH Terms: conditions — Bronchiolitis | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchiolitis children (Other): Under two years old patient with bronchiolitis will have thoracic radiology
  Interventions: Radiation: radiology

INTERVENTIONS:
Radiation: radiology — The investigators propose to performed a chest ultrasound in infants (<24 months) admitted for bronchiolitis with an available chest X-ray

SUMMARY:
The diagnosis of bronchiolitis, the most frequent lung infectious disease in infancy, is based on clinical examination. Chest X-ray is proposed when a lung parenchymal condensation is suspected. Chest ultrasound is supposed to be a useful tool in the diagnosis of these complication but is poorly evaluated. We aim to compare chest X-ray and chest ultrasound for the diagnosis of parenchymal condensation in infant with bronchiolitis.

DETAILED DESCRIPTION:
900 to 1000 children are admitted each year for bronchiolitis in the pediatric emergency department of the Toulouse Children Hospital. The diagnosis is based on clinical examination, but in some cases furthers examinations such as chest X-ray are necessary in order to look for a parenchymal condensation. Even if French recommendations do not place chest ultrasound in the care pathway to date, many recent studies show the usefulness, rapidity and reliability of ultrasound in parenchymal abnormalities. But regarding the bronchiolitis, few studies are available and including limited numbers of patients. In addition, the reduction of irradiation is a main goal, especially in children.

We propose to performed a chest ultrasound in infants (<24 months) admitted for bronchiolitis with an available chest X-ray, in order to compare the performance of both examinations (X-ray and ultrasound) for the diagnosis of parenchymal condensation. Besides, to correlate initial chest ultrasound results and clinical evolution, parents will be contacted by phone 1 month after inclusion.

Primary outcome: The primary outcome is the sensitivity and specificity values of chest ultrasound for the diagnosis of parenchymal condensations diagnosed by chest X-ray. Positive and negative predictive values will also be estimated. This outcome is evaluated at the first visit (T0).

Secondary outcomes:

* To describe chest X-ray and ultrasound abnormalities in bronchiolitis.
* To evaluate the performance of chest ultrasound to distinguish retractile and non-retractile opacities complicating bronchiolitis.
* To study the correlation between clinical evolution at 1-month (malaise, place and duration of hospitalization, re-hospitalization, oxygen therapy, antibiotic therapy) and chest ultrasound results.

Follow-up parameters are recorded during a telephone call 1 month after inclusion.

Study design : It is a longitudinal, monocentric and prospective study with the aim to evaluate a diagnostic examination.

ELIGIBILITY:
Inclusion Criteria:

* Two years old patient at emergency Hospital (CHU-Toulouse) for bronchiolitis and performing of thoracic radiology
* Informed consent formed to sign by family before the exam and the evidence of social security regime affiliation.

Exclusion Criteria:

* Patient with cardiopulmonary disease or underlying immunosuppression

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Presence of parenchymatous opacity | Inclusion
  Presence of parenchymatous opacity during thoracic radiological exam

SECONDARY OUTCOMES:
Radiological anomaly | Inclusion
  Description of all pleuropulmonary anomaly in every radiological anomaly
Parenchymatous retractable (or non retractable) opacity | Inclusion
  Assessment of radiographic capacity to differentiate Parenchymatous retractable (or non retractable) opacity

CONTACTS AND LOCATIONS:
Overall Officials: Marine MICHELET, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital des Enfants, Unité de pneumo-allergologie pédiatrique, Toulouse, France

IPD SHARING:
Plan to Share IPD: No